CLINICAL TRIAL: NCT03500614
Title: An Interventional Study on the Use of Air Cleaners to Mitigate Cardiopulmonary Health Impact of Indoor Exposure to Particles and Phthalates in Healthy Adults: a Randomized Double-blinded Crossover Trial.
Brief Title: The Use of Air Cleaners to Mitigate Cardiopulmonary Health Impact of Indoor Exposure to Particles and Phthalates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jing Huang, Assistant Professor, Peking University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2017095; 2017YFC0211601 (Other Grant/Funding Number: Ministry of Science and Technology of China); 2016YFC0207103 (Other Grant/Funding Number: Ministry of Science and Technology of China)
Record Dates: First submitted 2018-03-13; First posted 2018-04-18 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure; Lung Function; Inflammation; Oxidative Stress
Keywords: particulate matter; phthalates; cytokines; chemokines; epigenetics; DNA methylation; peripheral blood mononuclear cells; immune function
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants (n=57) will receive either true or sham air cleaner treatment for 1 week and then alternate the treatment after a wash out interval (Air cleaner use method 1). Exposure monitoring for PM2.5 will continue throughout the treatment period and air and fine particle phase phthalates samples will be collected during the last day (24 hours) of the treatment period; and health variables will be measured and biological samples will be collected immediately after the completion of each intervention period.
  Interventions: Behavioral: Air cleaner use method 1
- Cohort 2 (Experimental): Participants (n=32) will undergo extended treatment period covering the start, peak and end phases of smog episodes in Beijing, with either true or sham air cleaner treatment and then alternate the treatment after a wash out interval (Air cleaner use method 2). Exposure monitoring for PM2.5 will continue throughout the treatment period and repeated health examinations will be conducted at time points corresponding to the start, peak and end phases of the smog episodes.
  Interventions: Behavioral: Air cleaner use method 2

INTERVENTIONS:
Behavioral: Air cleaner use method 1 — All interventions in the first cohort will start at noon on Tuesday or Thursday and continue to the next morning of Tuesday or Thursday.
  Arms: Cohort 1
Behavioral: Air cleaner use method 2 — All interventions in the second cohort will start from the beginning to the end of smog episodes.
  Arms: Cohort 2

SUMMARY:
This study aims to evaluate whether a short-term intervention strategy using air cleaner reduces indoor exposure to airborne particles (particulate matter with an aerodynamic diameter ≤2.5μm, PM2.5) and phthalates and improves cardiopulmonary health among Chinese healthy adults based on a randomized double-blinded crossover trial.

DETAILED DESCRIPTION:
The randomized double-blind crossover trial includes two cohorts with different intervention and health examination settings and will be conducted in Beijing, China between November 2017-May 2018.

The first cohort plans to include 70 healthy college students who live in school dormitories, which were randomized into two dormitory groups to receive either true or sham air cleaner treatment for 1 week and then alternate the treatment after a wash out interval of at least 2 weeks (But in the enrollment, only 57 students were recruited actually). All participants and research staff are blinded to the group assignment. All participants are encouraged to stay in the dormitory with windows/doors tightly closed throughout the 1-week treatment period as far as possible, whereas necessary outdoor activities such as attending classes and dining in school canteens are allowed. All interventions will start at noon on Tuesday or Thursday and continue to the next morning of Tuesday or Thursday to avoid issues related to diurnal variation. Real-time PM2.5 concentrations will be measured using portable monitors and airborne PM2.5 mass samples will be collected in air filters throughout the treatment period. Air and fine particle phase phthalates samples will be collected using glass sampling tube filled with XAD2 macroporous resin and PM2.5 air filters respectively during the last day (24 hours) of the treatment period. Health variables, including blood pressure, lung function, fractional exhaled nitric oxide (FeNO), will be evaluated and biological samples including morning urine and fasting blood will be collected immediately after the completion of each treatment period. Efficacy of air cleaner treatment to reduce indoor exposure to particles and phthalates and related improvements in cardiopulmonary health variables will be evaluated using professional statistical methods.

The second cohort plans to include 30 healthy college students who will undergo extended treatment period covering the start, peak and end phases of smog episodes occurring in Beijing (To avoid dropout, 32 students were initially recruited). All interventions will start from the beginning to the end of typical smog episodes. PM2.5 exposure monitoring as detailed above will be performed throughout the treatment period and repeated health examinations will be conducted at time points corresponding to the start, peak and end phases of the smog episodes. Efficacy of air cleaner treatment to reduce indoor exposure to PM2.5 and related improvements in cardiopulmonary health variables throughout the smog episodes will be evaluated using professional statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy college students aged between 18 and 30 years old;
* Will stay within the central urban area of Beijing over the entire study including the wash-out period;
* BMI <30 kg/m3.

Exclusion Criteria:

* Current or ever smokers;
* A history of chronic respiratory diseases;
* A history of chronic cardiovascular diseases;
* Acute infections;
* Medication use in recent one month;
* Leave Beijing during the intervention.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure (BP) (cohort 1) | through the study completion, an average of 1-week
  The upper arm BP including both systolic pressure and diastolic pressure will be measured using an Omron J12 electronic sphygmomanometer for three times and the second and third readings will be used.
Lung function (cohort 1) | through the study completion, an average of 1-week
  Lung function measures including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and peak expiratory flow (PEF) will be determined using a Pony FX spirometer.
Fractional exhaled nitric oxide (FeNO) (cohort 1) | through the study completion, an average of 1-week
  FeNO levels will be measured using a portable NIOX VERO machine (Aerocrine AB, Solna, Sweden).
Urinary oxidative biomarkers (cohort 1) | through the study completion, an average of 1-week
  Morning urine samples will be collected and measured for malondialdehyde (MDA) and 8-iso-prostaglandinF2α (8-iso-PGF2α) using high performance liquid chromatography-mass spectrometry (HPLC-MS) and 8-hydroxydeoxyguanosine (8-OHdG) using enzyme linked immunosorbent assay (ELISA).
Circulating cytokine and chemokine biomarkers (cohort 1) | through the study completion, an average of 1-week
  Peripheral blood samples will be collected and measured for soluble CD40L(sCD40L), epidermal growth factor(EGF), Eotaxin-1, fibroblast growth factor 2(FGF2), fms-related tyrosine kinase 3 ligand(FLT3LG), Fractalkine, granulocyte-colony stimulating factor(G-CSF), granulocyte-macrophage colony-stimulating factor(GM-CSF), growth-related oncogene α(GROα), interferon-α2(IFN-α2), IFN-γ, interleukin-1α(IL-1α), IL-1β, IL-1R1, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p40, IL-12, IL-13, IL-15, IL-17, interferon-inducible protein-10(IP-10), monocyte chemoattractant protein-1(MCP-1), MCP-3, macrophage-derived chemokine(MDC), macrophage inflammatory protein-1α(MIP-1α), MIP-1β, platelet-derived growth factor-AA(PDGF-AA), PDGF-AB/BB, regulated upon activation normal T-cell expressed and secreted(RANTES), transforming growth factor-α(TGF-α), tumor necrosis factor-α(TNF-α), TNF-β and vascular endothelial growth factor(VEGF) using a liquid chip in Luminex platform.
Inflammatory and immune markers for peripheral blood mononuclear cell (PBMC) (cohort 1) | through the study completion, an average of 1-week
  The following inflammatory and immune markers of PBMC will be measured using labeled antibodies in multiplexed mass cytometry: p53, phospho-p53 (p-p53), p-mitogen-activated protein kinase 1/2 (pErk1/2), cell devision cycle protein 2 (cdc2), p-cdc2, signal transducer and activator of transcription 3 (STAT3), p-STAT3, serine/threonine kinase 1, ataxia telangiectasia mutated (ATM), p-ATM, p62, mammalian target of rapamycin (mTOR), p-mTOR, mitogen-activated protein kinases1+2, nuclear factor-kappa B p65 (NF-κB p65), p-NF-κB p65, c-Jun N-terminal kinase (JNK), p-JNK, glycoprotein 130 (gp130), p-gp130, Cyclin B1, p-Cyclin B1, phosphorylation protein kinase B, autophagy related gene 5, cluster differentiation antigen 4 (CD4), CD8, CD11c, CD14, CD20, CD56, toll-like receptor 4, myeloid differentiation primary response 88, TNF receptor associated factor 6, and interleukin-1 receptor-associated kinase 4.
Change in blood pressure from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  The upper arm BP including both systolic pressure and diastolic pressure will be measured using an Omron J12 electronic sphygmomanometer for three times and the second and third readings will be used.
Change in lung function from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  Lung function measures including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and peak expiratory flow (PEF) will be determined using a Pony FX spirometer.
Change in fractional exhaled nitric oxide (FeNO) from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  FeNO levels will be measured using a portable NIOX VERO machine (Aerocrine AB, Solna, Sweden).
Change in urinary oxidative biomarkers from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  Morning urine samples will be collected and measured for malondialdehyde (MDA) and 8-iso-prostaglandinF2α (8-iso-PGF2α) using high performance liquid chromatography-mass spectrometry (HPLC-MS) and 8-hydroxydeoxyguanosine (8-OHdG) using enzyme linked immunosorbent assay (ELISA).
Change in circulating cytokine and chemokine biomarkers from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  Peripheral blood samples will be collected and measured for soluble CD40L(sCD40L), epidermal growth factor(EGF), Eotaxin-1, fibroblast growth factor 2(FGF2), fms-related tyrosine kinase 3 ligand(FLT3LG), Fractalkine, granulocyte-colony stimulating factor(G-CSF), granulocyte-macrophage colony-stimulating factor(GM-CSF), growth-related oncogene α(GROα), interferon-α2(IFN-α2), IFN-γ, interleukin-1α(IL-1α), IL-1β, IL-1R1, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p40, IL-12, IL-13, IL-15, IL-17, interferon-inducible protein-10(IP-10), monocyte chemoattractant protein-1(MCP-1), MCP-3, macrophage-derived chemokine(MDC), macrophage inflammatory protein-1α(MIP-1α), MIP-1β, platelet-derived growth factor-AA(PDGF-AA), PDGF-AB/BB, regulated upon activation normal T-cell expressed and secreted(RANTES), transforming growth factor-α(TGF-α), tumor necrosis factor-α(TNF-α), TNF-β and vascular endothelial growth factor(VEGF) using a liquid chip in Luminex platform.

SECONDARY OUTCOMES:
DNA methylation (cohort 1) | through the study completion, an average of 1-week
  Genomic DNA methylation changes associated with indoor exposures will be screened using methylation chip in a group of selected participants and confirmed in both cohorts using bisulfite-polymerase chain reaction-pyrosequencing.
Concentrations of urinary phthalate metabolites (cohort 1） | through the study completion, an average of 1-week
  Fifteen main phthalate metabolites in morning urine samples including dimethyl phthalate (DMP), diethylphthalate (DEP), diisobuylphthalate (DIBP), dibutyl phthalate (DBP), bis(2-Methoxyethyl)phthalate (DMEP), bis(4-Methyl-2-pentyl)phthalate (DMPP), bis(2-Ethoxyethyl)phthalate (DEEP), dipentyl phthalate (DPP), dihexyl phthalate (DHP), benzyl butyl phthalate (BBP), bis(2-n-butoxyethyl)phthalate (DBEP), dicyclohexyl phthalate (DCHP), bis(2-Ethylhexyl)phthalate (DEHP), di-n-octyl phthalate (DnOP), dinonyl phthalate (DNP) will be quantified using gas chromatography-mass spectrometry (GC-MS).
Change in DNA methylation from baseline to during and after the intervention (cohort 2) | before, during and after the smog episodes (up to 10 days)
  Genomic DNA methylation changes associated with indoor exposures will be screened using methylation chip in a group of selected participants and confirmed in both cohorts using bisulfite-polymerase chain reaction-pyrosequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, PhD, Principal Investigator — Peking University; Shaowei Wu, PhD, Principal Investigator — Peking University
Locations (1):
- Department of Occupational & Environmental Health Sciences, School of Public Health, Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No